CLINICAL TRIAL: NCT05546918
Title: Users' Expectations and Co-design of a Digital Health Solution to Monitor Persisting Symptoms Related to COVID-19 Using Voice: a Mixed-methods Study
Brief Title: Co-design of a Digital Health Solution to Monitor Persisting Symptoms Related to COVID-19 Using Voice
Acronym: UpcomingVoice
Status: Completed | Type: Observational
Sponsor: Luxembourg Institute of Health (Other Government)
Responsible Party: Sponsor
Other Study IDs: UpcomingVoice
Record Dates: First submitted 2022-09-12; First posted 2022-09-21 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: COVID-19; Post-Acute COVID-19
Keywords: Post-Acute COVID-19; symptoms; vocal biomarkers; co-design; Digital health solution
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome | interventions — Surveys and Questionnaires; Interviews as Topic; Focus Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- People with Long COVID: Any people with persisting symptoms related to COVID-19 (With a Long COVID diagnosis or not)
  Interventions: Other: survey, interviews and focus groups
- Healthcare Professional: Healthcare professionals in charge of Long COVID patients
  Interventions: Other: survey, interviews and focus groups

INTERVENTIONS:
Other: survey, interviews and focus groups — The 2 groups of participants will be invited to:
  * complete an anonymous online survey
  * participate in individual semi-structured interviews and 2 focus groups

SUMMARY:
The UpcomingVoice project aims to co-design a digital health solution based on vocal biomarkers for screening and self-monitoring of frequently reported COVID-19-related symptoms with its end-users: 1) people with persisting COVID-19 related symptoms, with or without a Long COVID diagnosis and 2) healthcare professionals involved in the care of Long COVID patients.

To achieve this objective the UpcomingVoice study will determine:

* The needs, expectancies, acceptability, fears, barriers and leverages of the end-users regarding the use of voice to self-monitor or screen for Long COVID symptoms
* The specifications that such a mobile application should meet in order to be considered acceptable and effective by its intended users in terms of technological aspects (type of device, type of voice recordings…), frequency of utilisation, design etc.

The project consists in 2 separate parts : one anonymous online survey and one qualitative part based on semi-structured interviews and focus groups.

The results of this study will be the specifications of a voice-based digital health solution.

DETAILED DESCRIPTION:
The COVID-19 pandemic accelerated the use of remote patient monitoring in clinical practice or research for safety and emergency reasons, justifying the need for innovative digital health solutions to monitor key parameters or symptoms related to COVID-19 or Long COVID. A panel of experts from the National Institute for Health and Care Excellence (NICE) recommended the development of telemonitoring and encouraged self-management of acute and Long COVID symptoms in a tailored and accessible way for each patient.

Voice is an interesting approach to use for telemonitoring as it is easy-to-collect, quick, energy efficient, and inducing less burden for patients. To bring vocal biomarkers of different symptoms into clinical and real-life practice, they have to be implemented in a digital health solution, for example a smartphone application.

It is crucial to involve the end-users in the development of such a digital health solution and in this project involve them during the entire project course.

The study protocol, the participant's documents, and the questionnaires have been reviewed by both Long COVID patients and HCPs prior to submission.

The co-design process will consist in 3 steps, each involving both patients and HCPs:

* Step 1. An online survey to assess acceptability, expectancies and define the general specifications of the digital health solution based on vocal biomarkers
* Step 2. Individual interviews based on the results of the online survey, to deeply discuss the same themes than in the survey and to define the main specification of the solution
* Step 3. Focus groups to present prototypes of the digital health solution and to collect user's comments and suggestions At each step participants will receive feedback from the previous step. Finally, participants with Long COVID and HCPs willing to be deeply involved in our research will be invited to co-author the scientific article presenting the results of this research.

The project is based on a mixed methods study and will integrate both qualitative and quantitative methods. Participants will be invited to participate in:

1. Online anonymous survey 2 Online semi-structured individual interviews 3. Online Focus groups

ELIGIBILITY:
Inclusion Criteria:

* People with persisting symptoms related to COVID-19 (With Long COVID diagnosis or not) or Healthcare professional in charge of Long COVID patients
* Adults (>18 years)
* Male or female
* French speaking people

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participation in the study will be proposed to adults (men and women) with persisting COVID-19 related symptoms, with or without a Long COVID diagnosis and to healthcare professionals in charge of Long COVID patients.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-02-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of barriers and facilitators regarding the use of voice to self-monitor or screen for Long COVID symptoms | At baseline
  Specific questions will be asked in the online survey and during an individual online interview to identify the needs, expectancies, acceptability, fears, barriers and leverages regarding the use of voice as a monitoring tool
Definition of the specifications of a digital health solution based on vocal biomarkers to monitor and screen for COVID-19 related symptoms | At baseline
  Specific questions will be asked in the online survey, during an individual online interview and during focus groups regarding the main dimensions of a digital health solution (Engagement, functionality, aesthetics, information and general items ("Would you recommend", "Would you be interested in", etc..)

CONTACTS AND LOCATIONS:
Overall Officials: Aurelie FISCHER, MSc, Principal Investigator — Luxembourg Institute of Health
Locations (1):
- Luxembourg Institute of Health, Strassen, Luxembourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fagherazzi G, Fischer A, Ismael M, Despotovic V. Voice for Health: The Use of Vocal Biomarkers from Research to Clinical Practice. Digit Biomark. 2021 Apr 16;5(1):78-88. doi: 10.1159/000515346. eCollection 2021 Jan-Apr. PMID 34056518
- [Background] Fischer A, Zhang L, Elbeji A, Wilmes P, Oustric P, Staub T, Nazarov PV, Ollert M, Fagherazzi G. Long COVID Symptomatology After 12 Months and Its Impact on Quality of Life According to Initial Coronavirus Disease 2019 Disease Severity. Open Forum Infect Dis. 2022 Aug 5;9(8):ofac397. doi: 10.1093/ofid/ofac397. eCollection 2022 Aug. PMID 35983269
- [Background] Aguayo GA, Goetzinger C, Scibilia R, Fischer A, Seuring T, Tran VT, Ravaud P, Bereczky T, Huiart L, Fagherazzi G. Methods to Generate Innovative Research Ideas and Improve Patient and Public Involvement in Modern Epidemiological Research: Review, Patient Viewpoint, and Guidelines for Implementation of a Digital Cohort Study. J Med Internet Res. 2021 Dec 23;23(12):e25743. doi: 10.2196/25743. PMID 34941554
- [Derived] Fischer A, Aguayo GA, Oustric P, Morin L, Larche J, Benoy C, Fagherazzi G. Co-Design of a Voice-Based Digital Health Solution to Monitor Persisting Symptoms Related to COVID-19 (UpcomingVoice Study): Protocol for a Mixed Methods Study. JMIR Res Protoc. 2023 Jun 19;12:e46103. doi: 10.2196/46103. PMID 37335611